CLINICAL TRIAL: NCT01902329
Title: A Phase 1 Trial of SGN-CD33A in Patients With CD33-positive Acute Myeloid Leukemia
Brief Title: A Safety Study of SGN-CD33A in AML Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN33A-001
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Acute Myelogenous Leukemia; Acute Myeloid Leukemia; Acute Promyelocytic Leukemia
Keywords: Acute Myeloid Leukemia; Antibody-Drug Conjugate; CD33 Antigen; Immunotherapy; Drug Therapy; Acute Myelogenous Leukemia; Acute Promyelocytic Leukemia; APL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute | interventions — vadastuximab talirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SGN-CD33A + HMA (Experimental): SGN-CD33A with hypomethylating agent
  Interventions: Drug: HMA; Drug: SGN-CD33A
- SGN-CD33A Monotherapy (Experimental): SGN-CD33A
  Interventions: Drug: SGN-CD33A

INTERVENTIONS:
Drug: HMA — azacitidine 75 mg/m2 for 7 days or decitabine 20mg/m2 for 5 days
  Arms: SGN-CD33A + HMA
Drug: SGN-CD33A — Given intravenously on Day 1 or Days 1 and 4 every 3 weeks (SGN-CD33A Monotherapy) or given intravenously on the final HMA dosing day every 4 weeks (SGN-CD33A+HMA)
  Other Names: vadastuximab talirine

SUMMARY:
This study will examine the safety profile of vadastuximab talirine (SGN-CD33A) administered as a single agent and in combination with a hypomethylating agent (HMA). The main purpose of the study is to find the maximum tolerated dose (MTD, which is the highest dose that does not cause unacceptable side effects) of SGN-CD33A in patients with acute myeloid leukemia (AML). The MTD will be determined by observing the dose-limiting toxicities (the side effects that prevent further increases in dose) of SGN-CD33A. In addition, the pharmacokinetic profile and anti-leukemia activity of SGN-CD33A will be assessed.

DETAILED DESCRIPTION:
This study will explore SGN-CD33A as a monotherapy and in combination with a hypomethylating agent (HMA; i.e., azacitidine or decitabine). Initial study treatment with SGN-CD33A includes a maximum of 2 cycles of treatment for monotherapy and 4 cycles for combination cohorts. Patients who achieve documented CR or CRi (Monotherapy) or clinical benefit (Combination) during the first part of the study are eligible to continue treatment.

Additional monotherapy cohorts may include patients with relapsed acute promyelocytic leukemia, relapsed patients with nucleophosmin-1 gene mutation (absence of fms-like tyrosine kinase 3 mutation) (NPM1-mutated, FLT-3 wild type), alternate dosing schedules (fractionated dosing on Days 1 and 4), treatment naive patients with AML who declined intensive therapy, and patients who have relapsed after post-allogeneic stem cell transplant.

Patients in the combination cohort will be treated with azacitidine or decitabine per institutional practice prior to SGN-CD33A dosing. Expansion cohorts may be added for further evaluation of safety, pharmacokinetics, pharmacodynamics, and antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia, positive for CD33
* Eastern Cooperative Oncology Group status of 0 or 1
* Adequate baseline renal and hepatic function
* Central venous access
* Either achieved complete remission (greater than 12 weeks in duration) with initial induction/consolidation and have experienced relapse of disease or declined treatment with high-dose induction/consolidation
* Bone marrow blasts greater than or equal to 5% for relapsed patients, or greater than or equal to 20% for untreated patients

Exclusion Criteria:

* Inadequate lung function
* Prior allogeneic stem cell transplant, except for a specific cohort
* High-dose chemotherapy within 4 weeks of study drug
* Antileukemia treatment within 14 days of study drug (other than hydroxyurea or 6-mercaptopurine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03-18 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 1 month following last dose
Incidence of laboratory abnormalities | Through 1 month following last dose

SECONDARY OUTCOMES:
Blood concentrations of SGN-CD33A and metabolites | Through 3 weeks after dosing
Incidence of antitherapeutic antibodies | Through 1 month following last dose
Rate of complete remission | Up to 3 months
Duration of complete remission | Up to approximately 3 years
Relapse-free survival | Up to approximately 3 years
Overall survival | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Phoenix Ho, MD, Study Director — Seagen Inc.
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, The, Cleveland, Ohio
  - Charles A. Sammons Cancer Center / Baylor University Medical Center, Dallas, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Stein EM, Walter RB, Erba HP, Fathi AT, Advani AS, Lancet JE, Ravandi F, Kovacsovics T, DeAngelo DJ, Bixby D, Faderl S, Jillella AP, Ho PA, O'Meara MM, Zhao B, Biddle-Snead C, Stein AS. A phase 1 trial of vadastuximab talirine as monotherapy in patients with CD33-positive acute myeloid leukemia. Blood. 2018 Jan 25;131(4):387-396. doi: 10.1182/blood-2017-06-789800. Epub 2017 Dec 1. PMID 29196412